CLINICAL TRIAL: NCT01713738
Title: Open Label, Phase I/II Trial of Rituximab for Chronic, Severe Idiopathic Thrombocytopenic Purpura (ITP)in Children and Adolescents
Brief Title: Clinical Trial of Rituximab in Children and Adolescents With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neufeld, Ellis J, MD, PhD (Individual)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry); Glaser Pediatric Research Network (Network); Terrana ITP Research Fund (Other)
Responsible Party: Ellis J. Neufeld, MD, PhD, Children's Hospital Boston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHB 02-12-160; Genentec/IDEC U2591S; Glaser 435
Record Dates: First submitted 2012-10-18; First posted 2012-10-25 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Idiopathic Thrombocytopenic Purpura (ITP); Immune Thrombocytopenic Purpura (ITP)
Keywords: ITP; rituximab; bleeding score; platelet count; health-related quality of life; HRQL
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental)
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — infusion of 4 weekly doses of 375 mg/m2 rituximab

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of rituximab in children ages 18 months to 18 years, who have severe, chronic ITP. Eligible patients with either primary or secondary ITP are treated with rituximab once a week for 4 doses, and then followed for up to one year. Response is defined as having a platelet count greater than or equal to 50,000/mL on four consecutive weekly measures beginning anytime in weeks 9 - 12.

DETAILED DESCRIPTION:
The purpose of this open label, phase I/II study is to evaluate the safety and efficacy of rituximab in children ages 18 months to 18 years, who have severe, chronic ITP. Eligible patients with either primary or secondary ITP are treated with rituximab once a week for 4 doses, and then followed for up to one year. The primary and secondary objectives for safety and efficacy are as follows:

Primary

1. Efficacy: To evaluate the effectiveness of rituximab in severe or refractory pediatric ITP, with response defined as follows: platelet count greater than or equal to 50,000/mL on four consecutive weekly measures beginning anytime in weeks 9 - 12 (day 57 - day 84), with the first and fourth measure being spaced at least 22 days apart (i.e., once established during the 9 - 12 week timeframe, the response would be defined as beginning at the first one of these measures). All measurements must be independent of supportive care, as follows: 1) no IVIG (intravenous immunoglobulin) administration within 7 days of the first measure or at any time between measures, 2) no initiation of a 4-day corticosteroid "pulse" within 7 days of the first measure or at any time between measures, 3) no RHo (D) immunoglobulin (WinRHo-SDFTM ) administration within 7 days of the first measure or at any time between measures, and 4) no platelet transfusions administered within 7 days of the first measure or at any time between measures.
2. Safety: To obtain further safety information on rituximab in this clinical setting using Genentech standard safety monitoring and SAE reporting. In addition, the frequency of hypogammaglobulinemia will be assessed as the incidence of IgG levels <1/2 the lower limit of normal for age.

Secondary

1. To evaluate the one-year clinical course of severe or refractory ITP patients treated with a single course of rituximab. What fraction of responsive patients maintains this response?
2. To assess the need for salvage therapy (supportive care) in this severely affected group of patients during the clinical trial.
3. To evaluate the rate of "early response," defined as: platelets greater than or equal to 50,000/mL at least one week off rescue therapy, BEFORE day 57, and continuing for four consecutive weeks.
4. To follow the trend of bleeding scores from onset of therapy through the duration of the trial.
5. To assess the incidence of hypogammaglobulinemia requiring intervention (IgG level <1/2 of lower limit of normal for age) in this setting. IVIG 400 mg/kg monthly will be used to treat hypogammaglobulinemia.
6. To describe the health-related quality of life (HRQL) of children with severe or refractory ITP, based on parent report and to assess the impact on the family, using standardized questionnaires. This is a pilot-scale objective.

ELIGIBILITY:
Inclusion Criteria:

severe, chronic ITP, including refractory; at least 6 months from diagnosis for refractory; at least 12 months from diagnosis for severe; platelet counts <10,000/mm3 twice in past 3 months without bleeding; platelet counts <20,000/mm3 twice in past 3 months with bleeding

-

Exclusion Criteria:

ever had B or T cell neoplasm; HIV/AIDS; allergy to murine antibodies; treatment with investigational immunosuppressive strategies within past 3 months -

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2003-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
platelet levels | 9 - 12 weeks after 1st dose of rituximab
hypogammaglobulinemia | over one year

SECONDARY OUTCOMES:
fraction of responsive patients maintaining response over 1 year | week 52
assessment of need for salvage therapy | first 12 weeks of trial
rate of early response before day 57 | before day 57, and 4 additional weeks
trend of bleeding scores throughout trial | over one year
description of health-related quality of life | over one year

CONTACTS AND LOCATIONS:
Overall Officials: Ellis J Neufeld, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (9):
- United States (9):
  - UCLA, Mattel Children's Hospital, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Hospital Boston, Boston, Massachusetts
  - Van Eslander Cancer Center, St. John Hospital, Detroit, Michigan
  - Weill Medical College at Cornell University, New York, New York
  - Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas